CLINICAL TRIAL: NCT01978067
Title: Safety ,Validity and Quality of (Sexual)Life of Vaginal Operation in The Treatment Of Previous Cesarean Scar Defect
Brief Title: Quality of Life and Sexual Function of Vaginal Operation in The Treatment Of Previous Cesarean Scar Defect
Acronym: PCSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shu-Qin Chen (Other)
Responsible Party: Sponsor-Investigator, Shu-Qin Chen, associate professor of gynaecology and obstetricsf, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: CHEN-PCSD; PCSD-2013 (Other: Hospital Ethical Committee)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Quality of Life; Sexual Activity
Keywords: Uterine Scar From Previous Cesarean Delivery; previous caesarean scar deficiency; transvaginal resection; quality of life; sexual activity
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- transvaginal resection of Uterine Scar: transvaginal resection of Uterine Scar From Previous Cesarean Delivery
  Interventions: Procedure: transvaginal resection of Uterine Scar

INTERVENTIONS:
Procedure: transvaginal resection of Uterine Scar — Expose, grasp and traction the cervix. An incision was made at the anterior cervicovaginal junction, and the bladder was dissected away until the anterior peritoneal reflection was identified. The anterior drawing hook was inserted.into the vaginal incision to retract the bladder upwards. The PCSD was identified as a'fornix' located in the anterior part of the lower uterine segment. A transverse incision was made to remove the scar deficiency, and the edges of the incision were trimmed with scissors, and the myometrial and vaginal defects were closed.

SUMMARY:
The aim of this study is to further demonstrate the safety , validity and quality of (sexual)life of vaginal operation for previous cesarean scar defect resection.

DETAILED DESCRIPTION:
collect all the patients'clinical information,use two questionnaire (the HRQoL and FSFI)to estimate patients' general healthy and sexual function before surgery and postoperation in 1 month,3 months and 6 months

ELIGIBILITY:
Inclusion Criteria:

* preoperative diagnosed as PCSD
* hemodynamic stability

Exclusion Criteria:

* irregular menstrual cycle
* using IUD
* complicating other disease also causing vaginal bleeding,such as endometrial polyp,submucous myoma and functional uterine bleeding.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 patients diagnosed PCSD scheduled for vaginal operation in The First Affiliated Hospital between December 2013 and December 2015
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The safety of transvaginal resection of caesarean scar deficiency in the treatment of PCSD | one week
  blood loss, hemoglobin in the first postoperative day, operation time, preoperative and postoperative complications,change to other treatment,vaginal bleeding after surgery and length of stay are collected to evaluate the safety of this procedure.

SECONDARY OUTCOMES:
the effectiveness of transvaginal resection of caesarean scar deficiency in the treatment of PCSD. | one year
  Observation of menstruation in three months,six months and nine months after surgery is applied for evaluating the effectiveness of this procedure and transvaginal ultrasound,hysteroscopy and Gynecological Examination are performed after surgery.Situation of fertility ,(sex)quality of life after surgery also are very important indicator of this procedure effectiveness

OTHER OUTCOMES:
the result of transvaginal resection of caesarean scar deficiency in affecting quality of (sex)life. | one year
  two questionnaires results:FSFI and HRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Chen Shu-Qin, M.D&PhD, Study Director — First Affiliated Hospital, Sun Yat-Sen University; Yao Shu-Zhong, M.D&Ph.D, Study Chair — First Affiliated Hospital, Sun Yat-Sen University; Fan Li, M.D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China